CLINICAL TRIAL: NCT06577298
Title: A Phase I/II Randomized, Double-blind, Positive-controlled Dose-exploration Study to Evaluate the Safety and Immunogenicity of a Virus-like Particle (VLP) Based Vaccine Against Poliomyelitis (VLP-Polio) in Infants From 6 Weeks of Age and Toddlers 12-18 Months of Age
Brief Title: A Study to Evaluate the Safety and Immunogenicity of VLP-Polio in Infants and Toddlers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTP-VLP-002
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2024-08

CONDITIONS: Poliomyelitis
Keywords: Vaccine; Trivalent; Immunogenicity; Safety; 12-18 months toddlers; 2 months infants
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Phase I, Toddler Group A, Experimental vaccine, High dose, IM (Experimental): One dose of VLP-Polio on Day 0
  Interventions: Biological: VLP-Polio high dose
- Phase I, Toddler Group A, Control vaccine, IM (Active Comparator): One dose of IPV control on Day 0
  Interventions: Biological: Vaccine Poliomyelitis Inactivated (IPV)
- Phase I, Infant Group B, Experimental vaccine, Low-adjuvant dose, IM (Experimental): 4 dose of VLP-Polio on Day 0, Day 28, Day 56 and Month 12-18 of age
  Interventions: Biological: Recombinant Trivalent Poliomyelitis Vaccine (Sf-RVN Cell) (VLP-Polio) low adjuvant dose
- Phase I, Infant Group B, Control vaccine, IM (Active Comparator): 4 dose of IPV on Day 0, Day 28, Day 56 and Month 12-18 of age
  Interventions: Biological: Vaccine Poliomyelitis Inactivated (IPV)
- Phase I, Infant Group C, Experimental vaccine, Medium dose, IM (Experimental): 4 dose of VLP-Polio on Day 0, Day 28, Day 56 and Month 12-18 of age
  Interventions: Biological: VLP-Polio medium dose
- Phase I, Infant Group C, Control vaccine, IM (Active Comparator): 4 dose of IPV on Day 0, Day 28, Day 56 and Month 12-18 of age
  Interventions: Biological: Vaccine Poliomyelitis Inactivated (IPV)
- Phase I, Infant Group D, Experimental vaccine, High dose, IM (Experimental): 4 dose of VLP-Polio on Day 0, Day 28, Day 56 and Month 12-18 of age
  Interventions: Biological: VLP-Polio high dose
- Phase I, Infant Group D, Control vaccine, IM (Active Comparator): 4 dose of IPV on Day 0, Day 28, Day 56 and Month 12-18 of age
  Interventions: Biological: Vaccine Poliomyelitis Inactivated (IPV)
- Phase II, Infant Group E, Experimental vaccine, Low-adjuvant dose, IM (Experimental): 4 dose of VLP-Polio on Day 0, Day 28, Day 56 and Month 12-18 of age
  Interventions: Biological: Recombinant Trivalent Poliomyelitis Vaccine (Sf-RVN Cell) (VLP-Polio) low adjuvant dose
- Phase II, Infant Group E, Control vaccine, IM (Active Comparator): 4 dose of IPV vaccine on Day 0, Day 28, Day 56 and Month 12-18 of age
  Interventions: Biological: Vaccine Poliomyelitis Inactivated (IPV)
- Phase II, Infant Group F, Experimental vaccine, Medium dose, IM (Experimental): 4 dose of VLP-Polio on Day 0, Day 28, Day 56 and Month 12-18 of age
  Interventions: Biological: VLP-Polio medium dose
- Phase II, Infant Group F, Control vaccine, IM (Active Comparator): 4 dose of IPV on Day 0, Day 28, Day 56 and Month 12-18 of age
  Interventions: Biological: Vaccine Poliomyelitis Inactivated (IPV)
- Phase II, Infant Group G, Experimental vaccine, High dose, IM (Experimental): 4 dose of VLP-Polio on Day 0, Day 28, Day 56 and Month 12-18 of age
  Interventions: Biological: VLP-Polio high dose
- Phase II, Infant Group G, Control vaccine, IM (Active Comparator): 4 dose of IPV on Day 0, Day 28, Day 56 and Month 12-18 of age
  Interventions: Biological: Vaccine Poliomyelitis Inactivated (IPV)

INTERVENTIONS:
Biological: Recombinant Trivalent Poliomyelitis Vaccine (Sf-RVN Cell) (VLP-Polio) low adjuvant dose — 4 doses of VLP-Polio vaccine (0.5ml) at 2, 3, 4 months and 12-18 months of age for infants
  Arms: Phase I, Infant Group B, Experimental vaccine, Low-adjuvant dose, IM; Phase II, Infant Group E, Experimental vaccine, Low-adjuvant dose, IM
Biological: VLP-Polio medium dose — 4 doses of VLP-Polio vaccine (0.5ml) at 2, 3, 4 months and 12-18 months of age for infants
  Arms: Phase I, Infant Group C, Experimental vaccine, Medium dose, IM; Phase II, Infant Group F, Experimental vaccine, Medium dose, IM
Biological: VLP-Polio high dose — 1 dose of VLP-Polio vaccine (0.5ml) on day 0 for toddlers, 4 doses at 2, 3, 4 months and 12-18 months of age for infants
  Arms: Phase I, Infant Group D, Experimental vaccine, High dose, IM; Phase I, Toddler Group A, Experimental vaccine, High dose, IM; Phase II, Infant Group G, Experimental vaccine, High dose, IM
Biological: Vaccine Poliomyelitis Inactivated (IPV) — 1 dose of IPV vaccine (0.5ml) on day 0 for toddlers, 4 doses at 2, 3, 4 months and 12-18 months of age for infants
  Arms: Phase I, Infant Group B, Control vaccine, IM; Phase I, Infant Group C, Control vaccine, IM; Phase I, Infant Group D, Control vaccine, IM; Phase I, Toddler Group A, Control vaccine, IM; Phase II, Infant Group E, Control vaccine, IM; Phase II, Infant Group F, Control vaccine, IM; Phase II, Infant Group G, Control vaccine, IM

SUMMARY:
This is a phase I/II randomized, double-blind, and positive-controlled study. Participants in the phase I toddler group will receive 1 dose of either high dose VLP-Polio (Dose H) or control vaccine in a ratio of 3:1. The phase I infant cohort will have 4 arms randomly assigned to receive either investigational vaccine (Low-adjuvant dose VLP-Polio, Medium dose VLP-Polio, or High dose VLP-Polio or control vaccine in a ratio of 3:1. Phase II infant cohort will have 4 arms randomly assigned to receive either investigational vaccine (Low-adjuvant dose VLP-Polio, Medium dose VLP-Polio, or High dose VLP-Polio or control vaccine in a ratio of 3:1. Each infant participant will be administrated 3 doses of the assigned vaccine with 28 days apart, and the booster dose will be given when the infant is 12-18 months old. Enrollment of Phase I and Phase II will be staggered in descending order of age group but ascending order of dosing levels. Blood and mucosal samples will be collected for immunogenicity evaluation over the time course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy toddlers aged 12-18 months at the time of screening, and have completed primary immunization of polio vaccine according to the national government program in the first year of life.
* Healthy infants aged 6 weeks to 2 months (42 to 98 days, with the day of birth considered day of life 1), and who have not received any polio vaccines.
* Able to obtain written informed consent from parent(s) or legal guardian(s).
* Participants and their parents or legal guardian(s) can comply with trial procedures, are available for the duration of follow-up, and have a suitable telephone contact available.

Exclusion Criteria:

Exclusion criteria for the first dose:

* Current polio disease or history of polio disease.
* Toddlers who have an interval of less than 5 months since their last dose of the polio vaccine.
* Infants born at < 37 weeks of gestation.
* Children with a birth weight < 2500g and a body weight < 3500g at the time of enrollment.
* Body temperature ≥37.5°C (the visit may be rescheduled when this criterion is met).
* Have congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.
* Any moderate or severe acute illness.
* Any abnormal vital signs.
* History of epilepsy, convulsions, or parent with congenital cognitive disability, dementia, or intellectual disabilities.
* Have received immunosuppressive treatment, cytotoxic treatment, glucocorticoid treatment, etc. (excluding local treatment, surface treatment of acute non-concurrent dermatitis, or spray treatment of allergic rhinitis).
* Received or plan to receive blood/plasma products or immunoglobulins throughout the study period or prior to study vaccination.
* History of serious adverse events and/or severe allergic reactions (e.g., systemic allergic reactions) to any component of the study vaccine.
* History of known disturbance of coagulation or blood disorder that could cause anemia or excess bleeding (e.g., thalassemia, coagulation factor deficiencies, severe anemia at birth).
* Immunocompromised individuals with known or suspected immunodeficiency as determined by medical history and/or physical examination (e.g., history of pancreatic, liver, spleen, kidney disease or history of resection).
* Administration of other vaccines within 7 days.
* Participation in other interventional studies within 28 days prior to screening and/or during study participation.
* Household member or sibling who has received or is scheduled to receive OPV in the previous 3 months until 5 weeks after the third dose of the primary immunization series.
* The participant is a direct descendant (child or grandchild) of any person employed by the Sponsor, the contract research organization (CRO), the investigator, or study site personnel.
* History or current evidence of any condition or therapy which might confound the results of the study, interfere with the participant's participation for the full duration of the study, indicate suspected diseases, or is not in the best interest of the participants to participate, in the opinion of the treating investigator.
* Family history of any medical conditions, that in the investigating doctor's opinion, could affect the trial outcomes.
* Any reason or condition the investigator considers sufficient to make a participant ineligible for participation in the study.

Exclusion criteria for the subsequent doses:

* Severe allergic reaction after the previous vaccination.
* Serious adverse events caused by the previous vaccination.
* Newly identified symptoms or newly occurred cases after the first vaccination that do not meet the inclusion criteria for the first dose, or that meet the exclusion criteria for the first dose. The decision to discontinue participation is determined by the investigator.
* Other reasons for exclusion considered by the investigating doctor .

Ages: 6 Weeks to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Phase I: Percentage of participants with solicited adverse events (AEs) | Within 7 days after each vaccination
Phase II: Percentage of participants with solicited adverse events (AEs) | Within 7 days after each vaccination
Phase II: Seroconversion rate of neutralizing antibodies against Sabin and wild-type poliovirus type 1, 2, and 3 | Day 0 before vaccination and on Day 28 after the 3rd dose vaccination

SECONDARY OUTCOMES:
Phase I: Percentage of participants with unsolicited AEs | Within 28 days after each vaccination
Phase I: Percentage of participants with solicited AEs | Within 30 minutes after each vaccination
Phase I: Percentage of participants experiencing serious adverse events (SAEs) | Through study completion, Toddlers about 6 months, Infant about 20-22 months.
Phase I: Geometric mean titer (GMT) of neutralizing antibodies against Sabin and wild-type poliovirus type 1, 2, and 3 in toddlers | Day 0 before vaccination and on Day 28 after the vaccination
Phase I: Seroprotection rate of neutralizing antibodies against Sabin and wild-type poliovirus type 1, 2, and 3 in toddlers | Day 0 before vaccination and on Day 28 after the vaccination
Phase I: Seroconversion rate of neutralizing antibodies against Sabin and wild-type poliovirus type 1, 2, and 3 in toddlers | Day 0 before vaccination and on Day 28 after the vaccination
Phase I: GMT of neutralizing antibodies against Sabin and wild-type poliovirus type 1, 2, and 3 in infants | Day 0 before vaccination and on Day 28 after the 3rd dose vaccination
Phase I: Seroprotection rate of neutralizing antibodies against Sabin and wild-type poliovirus type 1, 2, and 3 in infants | Day 0 before vaccination and on Day 28 after the 3rd dose vaccination
Phase I: Seroconversion rate of neutralizing antibodies against Sabin and wild-type poliovirus type 1, 2, and 3 in infants | Day 0 before vaccination and on Day 28 after the 3rd dose vaccination
Phase II: Percentage of participants with unsolicited AEs | Within 28 days after each vaccination
Phase II: Percentage of participants with solicited AEs | Within 30 minutes after each vaccination
Phase II: Percentage of participants experiencing SAEs | Through study completion, Toddlers about 6 months, Infant about 20-22 months.
Phase II: GMT of neutralizing antibodies against Sabin and wild-type poliovirus type 1, 2, and 3 | Day 0 before vaccination and on Day 28 after the 3rd dose vaccination
Phase II: Seroprotection rate of neutralizing antibodies against Sabin and wild-type poliovirus type 1, 2, and 3 | Day 0 before vaccination and on Day 28 after the 3rd dose vaccination
Phase II: GMT of neutralizing antibodies against Sabin and wild-type poliovirus type 1, 2, and 3 in extended immunogenicity subgroup participants. | Month 6 after the 3rd dose vaccination
Phase II: Seroprotection rate of neutralizing antibodies against Sabin and wild-type poliovirus type 1, 2, and 3 in extended immunogenicity subgroup participants. | Month 6 after the 3rd dose vaccination
Phase II: Seroconversion rate of neutralizing antibodies against Sabin and wild-type poliovirus type 1, 2, and 3 in extended immunogenicity subgroup participants. | Month 6 after the 3rd dose vaccination

OTHER OUTCOMES:
Phase II: GMT of neutralizing antibodies against Sabin and wild-type poliovirus type 1, 2, and 3 in extended immunogenicity subgroup participants. | Day 0 before booster vaccination, on Day 28 and Month 6 after the booster vaccination
Phase II: Seroprotection rate of neutralizing antibodies against Sabin and wild-type poliovirus type 1, 2, and 3 in extended immunogenicity subgroup participants. | Day 0 before booster vaccination, on Day 28 and Month 6 after the booster vaccination
Phase II: Seroconversion rate of neutralizing antibodies against Sabin and wild-type poliovirus type 1, 2, and 3 in extended immunogenicity subgroup participants. | Day 0 before booster vaccination, on Day 28 and Month 6 after the booster vaccination
Phase II: GMT of poliovirus type-specific neutralizing and binding antibodies (IgA, IgG, IgM) in stool samples in extended immunogenicity subgroup participants | Day 0 before vaccination, on Day 14 and Day 28 after the 3rd dose vaccination, on Day 0 before the booster vaccination, on Day 14 and Day 28 after the booster vaccination
Phase II: GMI (geometric mean fold increase) of poliovirus type-specific neutralizing and binding antibodies (IgA, IgG, IgM) in stool samples in extended immunogenicity subgroup participants | Day 0 before vaccination, on Day 14 and Day 28 after the 3rd dose vaccination, on Day 0 before the booster vaccination, on Day 14 and Day 28 after the booster vaccination
Phase II: GMT of poliovirus type-specific neutralizing and binding antibodies (IgA, IgG, IgM) in nasal samples in extended immunogenicity subgroup participants | Day 0 before vaccination, on Day 14 and Day 28 after the 3rd dose vaccination, on Day 0 before the booster vaccination, on Day 14 and Day 28 after the booster vaccination
Phase II: GMI of poliovirus type-specific neutralizing and binding antibodies (IgA, IgG, IgM) in nasal samples in extended immunogenicity subgroup participants | Day 0 before vaccination, on Day 14 and Day 28 after the 3rd dose vaccination, on Day 0 before the booster vaccination, on Day 14 and Day 28 after the booster vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Nina Putri, Dr, Principal Investigator — Dr. Cipto Mangunkusumo Hospital
Locations (1):
- Dr. Cipto Mangunkusumo Hospital, Jakarta, Indonesia